CLINICAL TRIAL: NCT05413460
Title: Effect of Transcutaneous Electrical Acupoint Stimulation on Postoperative Complications After Cranial Endovascular Treatment
Brief Title: Acupoint Stimulation and Cranial Endovascular Treatment
Acronym: ASSET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhihong LU (Other)
Responsible Party: Sponsor-Investigator, Zhihong LU, Professor, Air Force Military Medical University, China
Organization: Air Force Military Medical University, China (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: XJH-A-20200730
Record Dates: First submitted 2022-05-25; First posted 2022-06-10 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Cerebral Aneurysm
Keywords: transcutaneous electrical acupoint stimulation; endovascular treatment
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All participants are placed with electrodes at acupoints. The stimulator is put in an opaque box.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transcutaneous electrical acupoint stimulation (Experimental): Electrodes are placed at acupoints and connected to the stimulator. Electrical stimulation is given during surgery.
  Interventions: Device: transcutaneous electrical acupoint stimulation
- Control (No Intervention): Electrodes are placed at acupoints and connected to the stimulator. But no stimulation is given during surgery.

INTERVENTIONS:
Device: transcutaneous electrical acupoint stimulation — Electrodes are placed at acupoints and connected to the stimulator. Electrical stimulation is given during surgery.
  Other Names: TEAS
  Arms: transcutaneous electrical acupoint stimulation

SUMMARY:
In this prospective randomized controlled trial, the subjects will be assigned to group transcutaneous electrical acupoint stimulation (TEAS) and group control (no intervention). The postoperative outcomes including NIHSS (National Institute of Health stroke scale) score, morbidity and mortality will be evaluated during hospital stay and by one year after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥18 years
2. patients scheduled for cranial endovascular treatment

Exclusion Criteria:

1. American Society of Anesthesiologists class Ⅲ or higher
2. Hunt-Hess class Ⅲ or higher
3. body mass index (BMI) < 18 kg/㎡ or > 30kg/㎡
4. large or giant cerebral aneurysms with diameters greater than 15mm and minor cerebral aneurysms with diameters less than 3mm
5. posterior circulation infarction
6. recurrence of an cerebral aneurysms after endovascular procedures or surgical clipping
7. severe abnormal coagulation function, severe liver and kidney function damage, or combined with heart and respiratory system failure
8. injury or infection of the skin around the acupoint area
9. participate in other clinical researchers within 3 months
10. history of neurological or psychiatric diseases
11. patients with implanted electrophysiological device
12. use of sedative or analgesics before surgery
13. patients with difficulty in communication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2022-07-26 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
number of patients with major in-hospital postoperative complications | from end of surgery to discharge from hospital, in an average of 7 days
  major complications include myocardial infarction, heart failure, respiratory failure, mechanical ventilation, cerebral infarction, delirium and coma

SECONDARY OUTCOMES:
mortality by 30 days after surgery | from end of surgery to 30 days after surgery, in a total of 30 days
mortality by 3 months after surgery | from end of surgery to 3 months after surgery, in a total of 3 months
number of patients with major postoperative complications by 3 months after surgery | from end of surgery to 3 months after surgery, in a total of 3 months
  major complications include myocardial infarction, heart failure, respiratory failure, mechanical ventilation, cerebral infarction, delirium and coma
mortality by 6 months after surgery | from end of surgery to 6 months after surgery, in a total of 6 months
number of patients with major postoperative complications by 6 months after surgery | from end of surgery to 6 months after surgery, in a total of 6 months
  major complications include myocardial infarction, heart failure, respiratory failure, mechanical ventilation, cerebral infarction, delirium and coma
duration of postoperative in-hospital stay | from end of surgery to discharge from hospital, in an average of 7 days
serum interleukin-6 level at the end of the surgery | at end of the surgery
serum tumor necrosis factor-α level at the end of the surgery | at end of the surgery
episodes of hypotension during surgery | from start of surgery to end of surgery, in an average of 2 hours
  hypotension is defined as mean arterial pressure decreased by more than 20% of the baseline and persisting more than 1 minute
Score of Mini-mental State Examination at 1 day after surgery | at 24h after the end of surgery
  A Mini-Mental State Examination (MMSE) is a set of 30 questions that doctors and other healthcare professionals commonly use to check for cognitive impairment (problems with thinking, communication, understanding and memory). MMSE is with a maximal score of 30. A higher score means better cognitive function.
Score of Mini-mental State Examination at 3 days after surgery | at 72h after the end of surgery
  A Mini-Mental State Examination (MMSE) is a set of 30 questions that doctors and other healthcare professionals commonly use to check for cognitive impairment (problems with thinking, communication, understanding and memory). MMSE is with a maximal score of 30. A higher score means better cognitive function.
visual analog scale of pain at 1 day after surgery | at 24h after the end of surgery
  visual analogue scale is a scale of 10cm, 0 is for no pain, 10 is for pain that can not be tolerated. The participant is asked to mark the scale of their pain
visual analog scale of pain at 3 days after surgery | at 72h after the end of surgery
  visual analogue scale is a scale of 10cm, 0 is for no pain, 10 is for pain that can not be tolerated. The participant is asked to mark the scale of their pain
Quality of recovery score at 3 days after surgery | at 72h after the end of surgery
  Quality of recovery-40 is a questionnaire consisted of 40 questions about the recovery of the patient. Higher score means better recovery.
Rankin's score at 3 days after surgery | at 72h after the end of surgery
  Rankin's score consists of class of 6 levels and is used for evaluation of neurologic function. Higher score means worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing hospital, Fourth military medical university, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dhillon PS, Butt W, Podlasek A, McConachie N, Lenthall R, Nair S, Malik L, Hewson DW, Bhogal P, Makalanda HLD, James MA, Dineen RA, England TJ. Association between anesthesia modality and clinical outcomes following endovascular stroke treatment in the extended time window. J Neurointerv Surg. 2023 May;15(5):478-482. doi: 10.1136/neurintsurg-2022-018846. Epub 2022 Apr 21. PMID 35450928
- [Background] Campbell D, Deng C, McBryde F, Billing R, Diprose WK, Short TG, Frampton C, Brew S, Barber PA; MASTERSTROKE Study Group. Protocol for the MAnagement of Systolic blood pressure during Thrombectomy by Endovascular Route for acute ischemic STROKE randomized clinical trial: The MASTERSTROKE trial. Int J Stroke. 2022 Aug;17(7):810-814. doi: 10.1177/17474930211059029. Epub 2021 Nov 22. PMID 34806930
- [Background] Samuels N, van de Graaf RA, van den Berg CAL, Uniken Venema SM, Bala K, van Doormaal PJ, van der Steen W, Witvoet E, Boiten J, den Hertog H, Schonewille WJ, Hofmeijer J, Schreuder F, Schreuder TAHCML, van der Worp HB, Roos YBWEM, Majoie CBLM, Burke JF, van Es ACGM, van der Lugt A, Roozenbeek B, Lingsma HF, Dippel DWJ; MR CLEAN Registry Investigators. Blood Pressure in the First 6 Hours Following Endovascular Treatment for Ischemic Stroke Is Associated With Outcome. Stroke. 2021 Nov;52(11):3514-3522. doi: 10.1161/STROKEAHA.120.033657. Epub 2021 Sep 20. PMID 34538090